CLINICAL TRIAL: NCT01118767
Title: Evaluation of a Computer-Based System Using Cell Phones for HIV People in Peru
Acronym: Cell-POS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Walter Curioso Vilchez, Universidad Peruana Cayetano Heredia, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01TW007896 (NIH); R01TW007896 (NIH)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: HIV; Adherence; Sexual Behavior; HIV Infections
Keywords: Adherence; Appointment; Cell Phone; Cellular Phone; Clinic; Computers; Controlled Clinical Trials, Randomized; HIV/AIDS; Health Informatics; Health behavior; Information Technology; Internet; Intervention; Medication; Patient Satisfaction; Patient Self-Report; Patients; Peru; Phone; Public Health; Public Health Informatics; Randomized; Randomized Controlled Clinical Trials; Randomized Controlled Trials; Research; Secondary Prevention; Self-Report; Sex Behavior; Sexual Behavior; Sexually Transmitted Diseases; Sexually Transmitted Infection; Survey Instrument; Surveys; Telephone; Telephone, Cellular; Text; Unprotected Sex; Viral Load result; Vulnerable Populations; WWW; anti-retroviral therapy; consumer informatics; evidence base; follow-up; medication adherence; medication compliance; randomization; randomized controlled study; randomized trial; randomly assigned; safer sex; treatment adherence; user centered design; web; world wide web
MeSH Terms: conditions — Sexual Behavior; HIV Infections; Acquired Immunodeficiency Syndrome; Health Behavior; Patient Satisfaction; Sexually Transmitted Diseases; Unsafe Sex; Medication Adherence; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cell phone intervention (Experimental): Participant receives short text messages
  Interventions: Other: Cell phone intervention
- Standard of care (No Intervention): Participant receives standard of care support but not short text messages

INTERVENTIONS:
Other: Cell phone intervention — Participant receives short text messages, including: antiretroviral reminders, clinic appointment reminders, and preventive/educational messages
  Arms: Cell phone intervention

SUMMARY:
The investigators propose to develop and evaluate a computer-based intervention using cell phones to enhance adherence to antiretroviral treatment (ART) and support of HIV transmission risk-reduction among adult HIV-positive patients in Peru.

DETAILED DESCRIPTION:
Adherence to ART is critical for treatment success at the individual level and to avoid the onset of resistant strains of HIV. In Peru, where ART has recently been introduced, adherence to HIV treatment has not yet been addressed properly. Innovative approaches using information technologies such as cell phones are needed to increase adherence to ART for people with HIV/AIDS. The specific aims of the study are to: 1) Conduct formative research to assess culturally-specific behavioral messages to be included in the computer-based system; 2) Develop and test an interactive computer-based system using cell phones to enhance adherence to ART and to deliver HIV transmission risk reduction messages; 3) Evaluate the impact of the system on antiretroviral adherence and sexual risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive healthy male or female aged greater than or equal to 18
* Currently on ART
* Patients with a mobile phone for their personal use (not shared)
* Patients who know how to retrieve read text messages on their mobile phone
* Signed and dated written informed consent prior to admission to the study

Exclusion Criteria:

* Patients whose clinical condition might have interfered with the study (e.g., deafness, serious mental illness, mental retardation)
* Patients unable to give their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2011-12-01 (Actual); Study Completion 2011-12-10 (Actual)

PRIMARY OUTCOMES:
Self-reported medication adherence | 12 months
HIV-1 viral load | 12 months

SECONDARY OUTCOMES:
CD4 | 12 months
Self-reported HIV transmission risk behaviors | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter H Curioso, MD, MPH, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (2):
- Peru (2):
  - Universidad Peruana Cayetano Heredia, Lima
  - Via Libre, Lima